CLINICAL TRIAL: NCT05305157
Title: National Evaluation of the Expectations of Experts in Forensic Odontology on Telemedicine
Brief Title: Telemedicine and Forensic Odontology
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL22_0080
Record Dates: First submitted 2022-03-22; First posted 2022-03-31 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Dental Caries
Keywords: Public Health; Forensic odontology; Telemedicine; Identification post mortem; dentist who is an forensic odontology expert; member of the AFIO or UIO
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Experts on forensic odontology: Experts on forensic odontology, members of AFIO (French Association of odontological identification) and UIO (Odontological identification Unit)

SUMMARY:
The aim of this study is to identify the expectations of experts in forensic odontology on telemedicine.

This study could improve, in multiple cases post mortem body identification.

DETAILED DESCRIPTION:
Experts in forensic odontology will have to complete a questionnaire that will reveal their expectations and knowledge on telemedicine.

ELIGIBILITY:
Inclusion criteria:

- Experts in forensic odontology members of the AFIO or UIO association

Exclusion criteria:

- Dentist who not practicing forensic odontology

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Experts in forensic odontology members of the AFIO or UIO association
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-07-01 (Estimated)

PRIMARY OUTCOMES:
Evaluate the knowledge | 1 day
  Evaluate the knowledge expectations on telemedicine among experts on forensic odontology
Evaluate the expectations | 1 day
  Evaluate the expectations on telemedicine among experts on forensic odontology

SECONDARY OUTCOMES:
Highlight the key points to work in legal teleodontology | 1 day
  Highlight the key points to work in legal teleodontology according to the expectations of experts

CONTACTS AND LOCATIONS:
Overall Officials: Camille INQUIMBERT, PhD, Study Director — University Hospital, Montpellier; Camille AMMOR, GRANDATI, resident, Principal Investigator — UH MONTPELLIER
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC